CLINICAL TRIAL: NCT06158100
Title: A Phase 1 Study of Venetoclax in Combination With Azacitidine (VEN/AZA) Followed by Donor Lymphocyte Infusion (DLI) for Patients With Very High-Risk Acute Myeloid Leukemia (AML) Undergoing Allogeneic Hematopoietic Cell Transplant (HCT)
Brief Title: Venetoclax in Combination With Azacitidine (VEN/AZA) Followed by Donor Lymphocyte Infusion (DLI) for Patients With Very High-Risk Acute Myeloid Leukemia (AML) Undergoing Allogeneic Hematopoietic Cell Transplant (HCT)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding Sponsor decision due to review of efficacy data from other trials involving investigational product.
Sponsor: Antonio M Jimenez Jimenez (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Antonio M Jimenez Jimenez, Associate Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20230190
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Hematopoietic Cell Transplant (HCT)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Intervention Model Description: Phase 1 dose escalation/de-escalation and dose expansion design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VEN/AZA Dose Escalation/De-Escalation Cohort (Experimental): Participants in this group will begin Venetoclax and Azacitidine (VEN/AZA) combination therapy between day +42 and day +100 following hematopoietic cell transplant (HCT) infusion. VEN/AZA combination therapy will be administered for up to six (6) cycles, followed by up to six (6) additional cycles of Venetoclax monotherapy in the absence of disease progression or unacceptable toxicity. Each cycle is 28 days.
  Participants may also receive donor lymphocyte infusions (DLI) at the discretion of the treating physician, if certain criteria are met.
  Participants will receive up to one year (12 cycles) of study therapy, followed by up to one year of follow-up. Total participation duration is up to two years.
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Biological: Donor Lymphocyte Infusion
- VEN/AZA Expansion Cohort (Experimental): Participants in this group will receive VEN/AZA therapy at the most appropriate dose determined in Part 1. Participants may also receive donor lymphocyte infusions (DLI) at the discretion of the treating physician, if certain criteria are met.
  Participants will receive up to one year (12 cycles) of study therapy, followed by up to one year of follow-up. Total participation duration is up to two years.
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Biological: Donor Lymphocyte Infusion

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be given orally (PO) at the assigned doses of 50 or 100 mg once daily for 7, 14 or 21 days starting at day 1 of each 28-day cycle, for up to 12 cycles.
  Other Names: Venclexta; Venclyxto
Drug: Azacitidine — Azacitidine will be administered at a dose of 20mg/m^2 once daily subcutaneously (SC) or intravenously (IV) for five days (Days 1-5) of each 28-day cycle.
  Other Names: Vidaza; Azadine
Biological: Donor Lymphocyte Infusion — Donor lymphocyte infusions (DLI) may be administered at the discretion of the treating physician, if certain criteria are met. Participants may receive up to three (3) infusions of donor lymphocytes (a type of white blood cell) at the following dose levels and study timepoints:
  * DLI 1: 1x10^6 cluster of differentiation 3+ (CD3+) cells/kg, after cycle 3
  * DLI 2: 5x10^6 CD3+ cells/kg, after cycle 5, if there is persistent MRD
  * DLI 3: 1x10^7 CD3+ cells/kg, after cycle 7, if there is persistent MRD.

SUMMARY:
The purpose of this study is to see the effects of an investigational combination treatment of venetoclax, azacitidine, and donor lymphocyte infusion (DLI) in patients with high-risk AML receiving allogeneic hematopoietic cell transplantation, and to assess if the combination treatment is well tolerated and prevents disease relapse after transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18-75.
2. Patients with a histologic diagnosis of AML in morphological remission (<5% bone marrow (BM) blasts) prior to allogeneic hematopoietic cell transplantation and very high-risk for relapse defined as: (i) Presence of measurable residual disease (MRD) by multicolor flow cytometry (MFC) prior to transplant and receiving a reduced intensity conditioning (RIC) or nonmyeloablative (NMA) regimen (ii) Presence of MRD by MFC at day +30 post-transplant (iii) All patients with monosomal karyotype (MK) and those with 17p/tumor protein p53 (TP53) mutated disease irrespective of MRD status and intensity of conditioning regimen.
3. Adequate hematopoietic recovery after HCT, defined as:

   * Absolute neutrophil count (ANC) >= 1 x 10^9/L without daily use of myeloid growth factors
   * Platelet count >= 50 x 10^9/L without platelet transfusion within 1 week
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
5. Serum creatinine =< 1.5 mg/dL or creatinine clearance greater or equal than 40 cc/min
6. Serum bilirubin =< 1.5 x upper limit of normal (ULN)
7. Aspartate transaminase (AST) or alanine transaminase (ALT) =< 2.5 x ULN
8. Alkaline phosphatase =< 2.5 x UL
9. Negative serum or urine pregnancy test for women with reproductive potential.
10. A negative donor-specific antibody (DSA) assay (i.e., Micro-Flow Imaging (MFI) <m3000) for recipients of any mismatched graft (including haploidentical) HCT.

Exclusion Criteria:

1. Active disease (>5% blasts or any evidence of extra-medullary disease) at the time of transplantation or at day +30
2. Active acute graft-versus-host disease (aGVHD) requiring systemic IST or history of aGVHD grade III or higher.
3. Active chronic GVHD requiring systemic immunosuppressive therapy (IST).
4. Active uncontrolled systemic fungal, bacterial, or viral infection
5. Known active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
6. Significant active cardiac disease within the previous 6 months, including: New York Heart Association (NYHA) class III or IV congestive heart failure. Unstable angina, angina requiring surgical or medical intervention, and/or myocardial infarction.
7. History of any other malignancy within 2 years prior to study entry, except for: adequately treated in situ carcinoma of the cervix or carcinoma in situ of breast; basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; previous malignancy confined and surgically resected (or treated with other modalities) with curative intent; myelodysplastic syndrome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 13 months
  The RP2D of VEN/AZA therapy will be determined as the maximum tolerated dose of study treatment as assessed by treating physician using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of Participants Experiencing Treatment-Related Toxicity | Up to 13 months
  The number of participants experiencing treatment-related toxicity. Toxicity is defined as including dose limiting toxicities (DLTs), serious adverse events (SAEs) and adverse events (AEs) in study participants after starting study therapy. Toxicity will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to 24 months
  Recurrence-free survival (RFS) is defined as the elapsed time measured in months between the treatment start date (Cycle 1 Day 1) and date of documented disease recurrence or death from any cause. Alive patients without recurrence will be censored at the date of last documentation of recurrence-free status.
Overall Survival (OS) | Up to 24 months
  Overall survival (OS) is defined as the elapsed time measured in months between the treatment start date (Cycle 1 Day 1) and date of death from any cause. Alive patients will be censored at the date last known to be alive.
Proportion of Participants with Treatment-Related Mortality (TRM) | 180 days
  Treatment-related Mortality (TRM) is defined as the proportion of participants that died after starting study therapy, during the time of observation and in the absence of disease progression.
Number of Participants with acute GVHD After Allogeneic Hematopoietic Cell Transplant (HCT) | Up to 180 days
  The number of participants with acute graft-versus-host disease (aGVHD) among study participants will be reported at +100 and +180 days post-allogeneic HCT.
Number of Participants with chronic GVHD After Allogeneic Hematopoietic Cell Transplant (HCT) | 1 year
  The number of participants with chronic graft-versus-host disease (cGVHD) among study participants will be reported at one (1) year post-allogeneic HCT.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio M Jimenez Jimenez, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No